CLINICAL TRIAL: NCT05177900
Title: Investigating the Use of an Interphase Gap in Biphasic Pulses in DBS for ET Patients
Brief Title: Interphase Gap in Biphasic Stimulation in DBS for ET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Myles Mc Laughlin (Other)
Responsible Party: Sponsor-Investigator, Myles Mc Laughlin, Assistant Professor, KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: s61020_IPG
Record Dates: First submitted 2021-12-02; First posted 2022-01-05 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: The patient will be allocated to the both arms in a cross-over design (no interphase gap and interphase gaps of different lenghts). The order of the pulses will be delivered in a random order, and with a double-blind design. Of all pulses, the therapeutic window will be assessed acutely (3 times per pulse shape).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biphasic pulse without interphase gap (Active Comparator)
  Interventions: Device: Study Tool Computer
- Biphasic pulse with interphase gap (Experimental)
  Interventions: Device: Study Tool Computer

INTERVENTIONS:
Device: Study Tool Computer — Nonconventional pulses delivered with custom-ware designed by Boston Scientific

SUMMARY:
Deep Brain Stimulation (DBS) is a well established therapy in medication-refractory essential tremor (ET). Since the inception of DBS, cathodic pulses are used. Recent work suggests that biphasic pulses influence the therapeutic window when compared to cathodic pulses, when tested acutely. Animal studies and work from cochlear implants, show that the use of an interphase gap, influences the generation of action potentials. In this study, the goal is to investigate the use of an interphase gap in biphasic pulses in DBS for ET patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential tremor treated with Vim-DBS
* Normal impedances of DBS circuit
* Signed written informed consent

Exclusion Criteria:

* Active psychiatric disease or active alcohol or drug abuse
* Dementia
* History of recurrent or unprovoked seizures
* Relevant comorbidities that influence objective clinical assessment
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Therapeutic threshold (mA) | During uptitration of the amplitude (entire process takes 3-4 minutes)
  Amplitude needed to elicit tremor arrest, expressed in milliamperes (mA)
Side effect threshold (mA) | During uptitration of the amplitude (entire process takes 3-4 minutes)
  Amplitude needed to elicit non-transient side effects, expressed in milliamperes (mA)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boogers A, Peeters J, Van Bogaert T, De Vloo P, Vandenberghe W, Nuttin B, Mc Laughlin M. Interphase Gaps in Symmetric Biphasic Pulses Reduce the Therapeutic Window in Ventral Intermediate Nucleus of the Thalamus-Deep Brain Stimulation for Essential Tremor. Neuromodulation. 2023 Dec;26(8):1699-1704. doi: 10.1016/j.neurom.2022.09.012. Epub 2022 Nov 18. PMID 36404213